CLINICAL TRIAL: NCT04903522
Title: Can the Affects Conveyed by Baroque Music and Its Rhetoric Reduce Anxiety in Patients With Major Depressive Disorder Associated With Anxiety Symptoms?
Brief Title: Can the Affects Conveyed by Baroque Music Reduce Anxiety in Patients With Major Depressive Disorder ?
Acronym: BARHEPSY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-CHITS-002; 2021-A00216-35 (Other: Id-RCB)
Record Dates: First submitted 2021-05-19; First posted 2021-05-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Musical intervention; Anxiety
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Depressive patients (Experimental): Patients suffering from major depressive disorder with anxiety symptoms
  Interventions: Behavioral: Baroque music listening

INTERVENTIONS:
Behavioral: Baroque music listening — Patients will listen to a 30-minute "musical path" of baroque pieces. Before and after this, anxiety, depression and consciousness fluidity will be evaluated thanks to different questionnaires

SUMMARY:
Major depressive disorder, or characterized depressive episode, is a common illness that limits psychosocial functioning and impairs quality of life. The initial goal of treatment for a major depressive episode is complete remission of depressive symptoms. The most commonly used treatments are antidepressants, psychotherapy or a combination of medication and psychotherapy.

Music therapy can be considered as one of the complementary therapies in the treatment of the characterized depressive episode and many studies have shown a beneficial effect of musical interventions, even of short duration, on depression and anxiety.

In depressive disorders, therapies such as hypnosis or phenomenological psychotherapies lead to modifications of consciousness during which the subject finds the means, notably non-reflexive and in the realm of the imaginary, to overcome anxiety.

Generally speaking, in the field of musical cognition, it is considered that music affects the emotions. Unfortunately this approach is often insufficiently refined in cognitive psychology since it is most generally interested in the 6 fundamental emotions: joy, anger, fear, sadness, surprise, disgust. However, during the Baroque period (end of the 16th and 17th centuries), various philosophers and musicians analyzed with great finesse not these fundamental emotions, but more precisely the passions, or "shocks of the soul", that is to say the affects in their great diversity. These affects or passions are thus at the center of Baroque musical composition.

In the Barhepsy project, it is suggested that listening to Baroque music, thanks to the rhetoric of the passions included in it, would allow the mobilization of the patients' affects and thus reduce their state of anxiety. During a follow-up consultation, the effects of a 30-minute "musical path" of baroque pieces will be evaluated, exemplifying the reduction of anxiety and the subsequent appeasement, on the conscious experience of subjects suffering from a characterized depressive state associated with anxious symptoms.

DETAILED DESCRIPTION:
Major depressive disorder or characterized depressive episode is a common illness that limits psychosocial functioning and impairs quality of life. In 2008, the WHO ranked major depression as the third leading cause of disease burden worldwide and predicts that the disease will become the leading cause by 2030.

The 5th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) defines a depressive episode as the presence of a sad mood and/or anhedonia (loss of interest or pleasure) lasting at least 15 days, variably associated with other symptoms (appetite disturbance, sleep disturbance, feelings of guilt and worthlessness...). It also defines as an additional characteristic of this illness, anxiety and more precisely anxiety distress, i.e. the presence of the feeling of being tense, the feeling of unusual agitation and the difficulty to concentrate due to worry or fear.

When treating a major depressive episode, the initial goal is complete remission of depressive symptoms. The most commonly used treatments are antidepressants, psychotherapy or a combination of medication and psychotherapy. Although these treatments are effective, some studies show a high rate of discontinuation and poor remission and the use of complementary and alternative medicine is increasing.

Music therapy can be considered as one of the complementary therapies in the treatment of the characterized depressive episode and many studies have shown a beneficial effect of musical interventions, even of short duration, on depression and anxiety. However, the nature of the effects of music remains mysterious, and even if psychometric scales are used, the body of research lacks explanations of what happens in these improvement processes. To seek an explanation, there are two strategies: either one focuses on using a psychophysiological approach (with physiological or biological measures), or one tries to approach the problem through the changes in mental processes (i.e., the content and structure of consciousness) associated with this enhancement. This is the choice made in the Barhepsy protocol.

The Barhepsy project is part of the research program "Sounds, Music, Therapies: SoMuThé" developed at the CNRS (UMR 7061 PRISM, Marseille). It is part of the current trend of non-medicinal therapies by focusing on the beneficial effects of music and sound therapy. SoMuThé is a project inspired by a philosophical current called phenomenology. It is interested in the general problematic of the therapeutic effects of sound and music, not from the point of view of neurophysiological or cognitive processes evaluated by means of brain imaging or cognitive psychology experiments, but in what happens in the structure and contents of the consciousness of the subjects who benefit from such therapies. It is therefore more of a comprehension approach than an explanatory one, aiming at describing the conscious experience of these subjects in its reflexive and pre-reflexive component, and thus at understanding how their flow of consciousness is reconfigured. In depressive pathologies, therapies such as hypnosis or phenomenological psychotherapies lead to modifications of consciousness during which the subject finds means, notably non-reflexive and in the domain of the imaginary, to overcome anxiety.

Generally speaking, in the field of musical cognition, it is considered that music affects the emotions. Unfortunately this approach is often insufficiently refined in cognitive psychology since it is most generally interested in the 6 fundamental emotions: joy, anger, fear, sadness, surprise, disgust. However, during the Baroque period (end of the 16th and 17th centuries), various philosophers and musicians analyzed with great finesse not these fundamental emotions, but more precisely the passions, or "shocks of the soul", that is to say the affects in their great diversity. These affects or passions are thus at the center of Baroque musical composition.

In the Barhepsy project, it is suggested that listening to Baroque music, thanks to the rhetoric of the passions included in it, would allow to mobilize the patients' affects and thus reduce their state of anxiety. During a follow-up consultation, the effects of a 30-minute "musical path" of baroque pieces will be evaluated, exemplifying the reduction of anxiety and the subsequent appeasement, on the conscious experience of subjects suffering from a characterized depressive state associated with anxious symptoms. To study the structure and metamorphoses of consciousness during the experience of listening to music, will be assessed in these patients :

* anxiety by means of the STAI (State-Trait Anxiety Inventory) scale of Spielberger et al., 1983 , and depression by the BDI (Beck Depression Inventory-II) scale of Beck et al., 1996. These two questionnaires will make it possible to qualify (and quantify) these two clinical signs;
* the fluidity of consciousness by means of the EQFC scale. Indeed, consciousness is made more "fluid", less rigid after certain psychotherapies such as hypnosis.
* the reflexive and pre-reflexive contents of consciousness that can be obtained through experiential phenomenological interviews (EPE), which are based on guided introspection and allow the description of background experiences of consciousness.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over the age of 18
* Depressive state characterized by the DSM-V criteria
* Able to express his/her consent prior to participation in the study
* Affiliated to or beneficiary of a social security regimen

Exclusion Criteria:

* Deafness
* Suspected or diagnosed neurodegenerative disorder or other associated neurological pathology
* Comorbid psychotic disorder
* Pregnant women
* Patient under judicial protection (guardianship, curatorship...) or safeguard of justice
* Any other reason that, in the opinion of the investigator, would interfere with the evaluation of the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Anxiety assessed by State Trait Anxiety Inventory questionnaire | 1 day
  the minimum value is 20 and the maximum value is 80. Higher scores mean a worse outcome, high level of anxiety.

SECONDARY OUTCOMES:
Qualitative assessment scale of the fluency of consciousness (EQFC) | 1 day
  For State EQFC : the minimum value is 17 and the maximum value is 68. Higher scores mean a better outcome, high level of fluency. For "Trait" EQFC : the minimum value is 17 and the maximum value is 102. Higher scores mean a better outcome, high level of fluency.
Experiential phenomenological interviews (EPE) | 1 day
  based on guided introspection and allow the description of background experiences of consciousness
Depression assessed by Beck Depression Inventory-Second Edition (BDI-II) questionnaire | 1 day
  the minimum value is 0 and the maximum value is 63. Higher scores mean a worse outcome, high level of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Dias Alves, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (1):
- Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No